CLINICAL TRIAL: NCT02809274
Title: Incidence of Iron Deficiency in Polycythemia Vera (PV) and Association With Disease Features
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Meir Medical Center (Other)
Responsible Party: Principal Investigator, NOA LAVI md, Dr., Rambam Health Care Campus
Other Study IDs: 0186-16 CTIL
Record Dates: First submitted 2016-06-18; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Polycythemia Vera
Keywords: iron deficiency; polycythemia vera
MeSH Terms: conditions — Polycythemia Vera; Iron Deficiencies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum blood sample for hepcidin
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with PV, not newly diagnosed: Patients with clinically overt PV treated with watchful waiting (with or without aspirin), Phlebotomy (PHL), Hydrea or any other treatment.
  Influence of iron parameters on Patient-reported symptoms will be evaluated by questionnaires Blood serum samples will be taken for iron parameters analysis
  Interventions: Other: questionnaires
- Newly diagnosed patients with PV: Patients with clinically overt PV, newly diagnosed, before any treatment and before phlebotomy initiation.
  Influence of iron parameters on Patient-reported symptoms will be evaluated by questionnaires Blood serum samples will be taken for iron parameters analysis
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — • Influence of iron parameters on Patient-reported symptoms as assessed by Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) for assessment of the severity of symptoms, Quality of life evaluation by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and fatigue assessment by PROMIS Fatigue Scale: Short Form

SUMMARY:
Iron deficiency is a known feature of PV, occurs because of accelerated erythropoiesis, gastrointestinal blood loss and phlebotomy. Incidence and effect of iron deficiency in these patients is not well characterized. The study will assess the incidence of iron deficiency at diagnosis and during the course of PV, assess effect of iron deficiency on patient symptoms and its correlation with disease features.

This is a multicenter, non-interventional, non-randomized, prospective, observational study in an adult population (patients >18 years old) of patients who have been diagnosed with PV and are being followed in either community or academic medical centers in Israel.

DETAILED DESCRIPTION:
Background:

Within intestinal epithelial cells, some of the imported iron is incorporated into ferritin and other storage forms. A fraction of the iron taken up from the intestinal lumen passes through the cell, and is exported across the basolateral membrane to enter the body. Ferroportin, a metal ion transporter, serves as the basolateral iron exporter. Hepcidin regulates basolateral iron export by binding to ferroportin to trigger its internalization and lysosomal degradation. Each day, normal adults need 25 mg of iron to support hemoglobin production in maturing erythrocytes. This amount is much greater than the iron absorbed daily through the intestine. Obviously, iron needed for erythropoiesis must be acquired from supplies already existing in the body. The primary source of plasma iron is the reticuloendothelial macrophage system, which recovers iron from senescent and damaged erythrocytes. Other significant site of iron exchange is the liver.

Dietary iron absorption is enhanced in response to insufficient iron stores, increased erythropoietic demand or hypoxia. It is diminished in response to iron surfeit and inflammation. Based on these observations, four different "regulators" have been defined functionally: 1) The stores regulator modulates absorption several fold, increasing it in iron deficiency and decreasing it in iron overload. 2) The erythroid regulator is more potent-it can increase iron absorption 6- to 10-fold when erythropoiesis becomes iron -restricted, result either from iron deficiency or from accelerated production of erythroid precursors. 3) The hypoxia regulator mediates an increase in iron absorption in response to hypoxia, to allow for production of hemoproteins that bind and carry oxygen. 4) An inflammatory regulator also exists, which acts to decrease iron absorption in response to inflammation. All of these regulators act through a common, humoral effector that coordinates intestinal iron absorption and macrophage iron recycling. Hepcidin plays a major role in iron metabolism. It is produced in the liver, cleaved from a larger precursor molecule and secreted into the plasma. Circulating hepcidin attaches to ferroportin expressed on enterocytes and macrophages, causing ferroportin to be internalized into the cell and degraded in lysosomes. Hepcidin is induced in response to iron overload and inflammation. It is turned off in response to iron deficiency , ineffective erythropoiesis and hypoxia.

Polycythemia vera (PV) is one of the myeloproliferative neoplasms (MPNs) and is characterized by marrow hyperplasia with an increased number of erythrocytes, leukocytes and platelets in peripheral blood. Several studies have shown that iron deficiency is common in PV patients and can significantly influence the quality of their life. These complications are a result of expansive erythropoiesis, in addition to phlebotomy and/or gastrointestinal bleedings. The role of JAK2V617F in pathogenesis of iron deficiency in PV is also very intriguing. Kinase JAK2 is involved in signal transduction via the erythropoietin receptor. EPO is one of the hepcidin synthesis regulators. Some of the data has confirmed that JAK2 mutation may be involved in the regulation of the iron status in myeloproliferative disorders.

There are several reports in the literature on thrombotic complications in iron-deficient adults. Secondary thrombocytosis has been implicated in many cases.

In addition to the increased thrombotic risk associated with high platelet count, the decrease in antioxidant defense in iron deficiency may cause increased oxidant stress, which in turn may result in a tendency toward platelet aggregation. The abnormal platelet count and function observed in iron deficiency anemia could act synergistically to promote thrombus formation. Iron deficiency may contribute to a hypercoagulable state by affecting blood flow patterns within the vessels because of reduced deformability and increased viscosity of microcytic red blood cell.

Purpose:

Incidence and effect of iron deficiency in patients with PV is not well characterized. The study will assess the incidence of iron deficiency at diagnosis and during the course of PV, assess effect of iron deficiency on patient symptoms and its correlation with disease features.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of Polycythemia Vera (PV)
* Willing and able to provide written informed consent
* Willing and able to complete patient assessment questionnaires either alone or with minimal assistance from a caregiver and/or trained site personnel
* Under the supervision of a physician for the current care of PV including but not limited to watchful waiting, acetylsalicylic acid (ASA) 81mg or greater, antithrombotic therapy, Phlebotomy (PHL), Hydroxyurea (HU), interferon (recombinant or pegylated), busulfan, anagrelide

Exclusion Criteria:

* Diagnosis of myelofibrosis (MF) [including primary MF, post-PV MF, or post-essential thrombocythemia MF (post-ET MF)]
* Diagnosis of secondary Acute Myeloid Leukemia (AML)
* Diagnosis of Myelodysplastic Syndrome (MDS)
* Splenectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An adult population (patients >18 years old) of men and women who have been diagnosed with clinically overt PV will be enrolled. Sites will include both community and academic centers across Isreal.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of iron deficiency in patients with PV | 2 years

SECONDARY OUTCOMES:
Association between iron deficiency and other clinical features | 2 years
Influence of therapy (phlebotomies, hydroxyurea, other therapies) on iron parameters | 2 years
Influence of iron parameters on Patient-reported symptoms | 2 years
Influence of iron deficiency on arterial and venous thrombosis rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noa Lavi, Dr, Principal Investigator — Rambam Health Care Campus
Locations (12):
- Israel (12):
  - Emek Medical center, Afula
  - Soroka medical center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Bnei Zion medical center, Haifa
  - Rambam Medical center, Haifa
  - Meir Medical center, Kfar Saba
  - Sheba medical center, Ramat Gan
  - Kaplan medical center, Rehovot
  - Ziv Medical center, Safed
  - Maccabi, Tel Aviv
  - Tel Aviv Sourasky, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson TC, Grimes AJ, Slater NG, Wetherley-Mein G. Viscosity and iron deficiency in treated polycythaemia. Br J Haematol. 1981 Sep;49(1):123-7. doi: 10.1111/j.1365-2141.1981.tb07205.x. PMID 7272225
- [Background] Hutton RD. The effect of iron deficiency on whole blood viscosity in polycythaemic patients. Br J Haematol. 1979 Oct;43(2):191-9. doi: 10.1111/j.1365-2141.1979.tb03741.x. PMID 508628
- [Background] Kwapisz J, Zekanowska E, Jasiniewska J. Decreased serum prohepcidin concentration in patients with polycythemia vera. J Zhejiang Univ Sci B. 2009 Nov;10(11):791-5. doi: 10.1631/jzus.B0920217. PMID 19882752
- [Background] Rector WG Jr, Fortuin NJ, Conley CL. Non-hematologic effects of chronic iron deficiency. A study of patients with polycythemia vera treated solely with venesections. Medicine (Baltimore). 1982 Nov;61(6):382-9. doi: 10.1097/00005792-198211000-00004. No abstract available. PMID 7144531
- [Background] Franchini M, Targher G, Montagnana M, Lippi G. Iron and thrombosis. Ann Hematol. 2008 Mar;87(3):167-73. doi: 10.1007/s00277-007-0416-1. Epub 2007 Dec 8. PMID 18066546
- [Background] Birgegard G, Carlsson M, Sandhagen B, Mannting F. Does iron deficiency in treated polycythemia vera affect whole blood viscosity? Acta Med Scand. 1984;216(2):165-9. doi: 10.1111/j.0954-6820.1984.tb03788.x. PMID 6496176